CLINICAL TRIAL: NCT03898258
Title: Evaluation of the German Short-Form Qualiveen Questionnaire
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2019-07
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neurogenic bladder: individuals with chronic (≥12 months) neurogenic lower urinary tract dysfunction due to spinal cord injury (SCI)
  Interventions: Other: Qualiveen full version; Other: Qualiveen short-form

INTERVENTIONS:
Other: Qualiveen full version — Qualiveen full version questionnaire with 40 questions for assessing the quality of life in relation to bladder dysfunction in persons with neurogenic bladder
Other: Qualiveen short-form — Qualiveen short-form questionnaire with 8 questions for assessing the quality of life in relation to bladder dysfunction in persons with neurogenic bladder

SUMMARY:
Two questionnaires (Qualiveen full version and Qualiveen short-form (SF)), the project information and the consent form will be sent to individuals who are scheduled for an annual control at the urological out-patient clinic of the Swiss Paraplegic Centre and who fulfill the inclusion criteria. The patients will be asked to complete the two questionnaires and to bring the completed questionnaires and the signed consent form to the annual control at the Swiss Paraplegic Centre. Participants who have consented and completed the two questionnaires will receive the two questionnaires a second time 14 days later.

The primary objective of this project is to validate the German version of the SF Qualiveen questionnaire. The secondary objective is to evaluate the measurement properties of the German SF Qualiveen questionnaire in comparison with the full version.

ELIGIBILITY:
Inclusion Criteria:

* chronic (≥ 12 months) neurogenic lower urinary tract dysfunction due to SCI
* age ≥ 18 years

Exclusion Criteria:

* no informed consent as documented by signature
* history of concomitant neurological or psychological illness
* history of cognitive impairment
* insufficient German language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with chronic (≥ 12 months) neurogenic lower urinary tract dysfunction due to SCI
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
total score | baseline
  Total score of the Qualiveen questionnaire is the arithmetic mean of the four sub-scores. The sub-scores are assessed using a five-point Likert scale (minimum score 0, maximum score 4). The total score indicates how much quality of life is affected by bladder problems. The higher the score the more quality of life is affected.

SECONDARY OUTCOMES:
bother with limitations score | baseline
  Score of the domain bother with limitations of the Qualiveen questionnaire assessed with five-point Likert scale (minimum score 0, maximum score 4).The score indicates how much limitations due to bladder problems bother the affected individual. The higher the score the more the affected individuals are bothered.
change in bother with limitations score | baseline; 14 days
  Score of the domain bother with limitations of the Qualiveen questionnaire assessed with five-point Likert scale (minimum score 0, maximum score 4).The score indicates how much limitations due to bladder problems bother the affected individual. The higher the score the more the affected individuals are bothered
frequency of limitations score | baseline
  Score of the domain frequency of limitations of the Qualiveen questionnaire assessed with five-point Likert scale (minimum score 0, maximum score 4).The score indicates how often affected individuals experience limitations due to bladder problems. The higher the score the more often the affected individuals experience limitations due to bladder problems.
change in frequency of limitations score | baseline; 14 days
  Score of the domain frequency of limitations of the Qualiveen questionnaire assessed with five-point Likert scale (minimum score 0, maximum score 4).The score indicates how often affected individuals experience limitations due to bladder problems. The higher the score the more often the affected individuals experience limitations due to bladder problems.
fears score | baseline
  Score of the domain fears of the Qualiveen questionnaire assessed with five-point Likert scale (minimum score 0, maximum score 4).The score indicates how much fear due to bladder problems the affected individuals experience. The higher the score the more fear the affected individuals experience
change in fears score | baseline; 14 days
  Score of the domain fears of the Qualiveen questionnaire assessed with five-point Likert scale (minimum score 0, maximum score 4).The score indicates how much fear due to bladder problems the affected individuals experience. The higher the score the more fear the affected individuals experience
feelings score | baseline
  Score of the domain feelings of the Qualiveen questionnaire assessed with five-point Likert scale (minimum score 0, maximum score 4).The score indicates how much feelings are affected by bladder problems. The higher the score the more the feelings are affected.
change in feelings score | baseline; 14 days
  Score of the domain feelings of the Qualiveen questionnaire assessed with five-point Likert scale (minimum score 0, maximum score 4).The score indicates how much feelings are affected by bladder problems. The higher the score the more the feelings are affected.

OTHER OUTCOMES:
age (years) | baseline
gender | baseline
bladder evacuation method | baseline
  type of bladder evacuation method (e.g. intermittent catheterization) as reported by study participant
number of daily bladder evacuations (n/24h) | baseline
  how often does study participant empty bladder during 24h
urinary incontinence | baseline
  presence of urinary incontinence as reported by study participant

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Pannek, Prof, Principal Investigator — Schweizer Paraplegiker-Zentrum Nottwil
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No